CLINICAL TRIAL: NCT06247007
Title: Modulation of Host Inflammatory Response With Electro Acupuncture as an Adjunct to Non-Surgical Periodontal Therapy: A Randomized Clinical Trial
Brief Title: Electroacupuncture as an Adjunct to Non-Surgical Periodontal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Didem OZKAL EMINOGLU (Other)
Collaborators: Ataturk University (Other); The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Didem OZKAL EMINOGLU, assistant professor, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024/ EA
Record Dates: First submitted 2024-01-29; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Periodontal Diseases; Periodontal Inflammation; Periodontitis; Acupuncture; Electroacupuncture; Periodontal Pocket
Keywords: periodontitis; Acupuncture; Electroacupuncture; IL-6; IL-10; TNF-α; Cytokine; non-surgical periodontal therapy
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Periodontal Pocket | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EA (electroacupuncture) (Experimental): Individuals who underwent electroacupuncture addition to non-surgical periodontal therapy
  Interventions: Procedure: Electroacupuncture
- Control (No Intervention): Individuals who have non-surgical periodontal therapy only

INTERVENTIONS:
Procedure: Electroacupuncture — LI-4, LI-11, GV-14, GV-20 acupuncture points were needled bilaterally.
  Arms: EA (electroacupuncture)

SUMMARY:
The aim of this randomized, single-masked, controlled clinical trial study was to determine if the administration of electro acupuncture improves the outcomes obtained in combination with non-surgical periodontal therapy.

Participants will get non-surgical periodontal therap with/without electro acupuncture.

Researchers will compare EA and control groups to see if there is any relationship between acupuncture application clinical periodontal parameters,serum and saliva cytokine levels.

DETAILED DESCRIPTION:
Periodontitis is a prevalent complex chronic inflammatory oral disease that can result in the progressive destruction of tooth supporting tissues and eventual loss of teeth. Although pathogenic bacteria are the triggers and provokers of periodontal inflammation, the main determinant of the destruction is the host immunoinflammatory response. The host response is modified by many genetic and environmental factors as well as various systemic diseases.

Electroacupuncture (EA) has effects on both the immune system and inflammatory processes. The effect of acupuncture on the regulation of cytokine production has been mentioned in the literature. .

No study has been found in the literature about the effects of EA on the host modulation in periodontitis patients. In this study, the investigators aimed to examine the effect of electroacupuncture application on the host modulation at periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* absence of any systemic disease,
* pregnancy or breast feeding;
* not receiving anti-inflammatory drug therapy in the last 6 months, chemotherapy or radiotherapy;

Exclusion Criteria:

* Having a systemic disease such as cardiovascular, diabetes, hypertension, thyroid organ pathologies, chronic kidney failure
* pregnant/breastfeeding
* medication for any reason
* smoker/tobacco user
* other periodontal disease other than periodontitis
* chronic inflammatory disease (COPD, asthma)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Clinical periodontal parameters / clinical attachment level (CAL) | Baseline-week 3
  CAL was measured as the distance between the deepest point of the sulcus and the cemento-enamel junction
Clinical periodontal parameters / probing pocket depth (PPD) | Baseline-week 3
  PPD was measured as the distance between the deepest point of the sulcus and the gingival margin
Clinical periodontal parameters / bleeding on probing (BOP) | Baseline-week 3
  The presence of bleeding on probing is considered an objective sign of periodontal inflammation
Clinical periodontal parameters / plaque index (PI) | Baseline-week 3
  The amount of plaque present on the teeth was assessed using a plaque staining agent and graded according to the plaque index system
Clinical periodontal parameters / gingival index (GI) | Baseline-week 3
  The presence and extent of gingival inflammation and bleeding were graded according to the gingival index system
Biochemical findings | Baseline-day 7-week 3
  IL-6, IL-10, TNF-α

CONTACTS AND LOCATIONS:
Overall Officials: DİDEM ÖZKAL EMİNOĞLU, Study Director — Ataturk University
Locations (1):
- Atatürk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No